CLINICAL TRIAL: NCT00060476
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Evaluate the Effects of Rofecoxib in Decreasing the Risk of Prostate Cancer (ViP Study)
Brief Title: Treatment With MK0966 for the Prevention of Prostate Cancer (0966-201)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0966-201; Formally-P30A03LD; MK0966-201; 2006_414
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — rofecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: rofecoxib
  Other Names: MK0966
Drug: Comparator: placebo (unspecified)

SUMMARY:
To determine the efficacy and safety of an investigational compound (MK0966) for the prevention of prostate cancer.

DETAILED DESCRIPTION:
The duration of treatment is 6 years.

ELIGIBILITY:
Regular PSA testing and study biopsies required.

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15000 (Actual)
Dates: Start 2003-01-08 (Actual); Primary Completion 2004-12-08 (Actual); Study Completion 2004-12-08 (Actual)

PRIMARY OUTCOMES:
Time to prostate cancer | Duration of Treatment

SECONDARY OUTCOMES:
Time to aggressive prostate cancer | Duration of Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] van Adelsberg J, Gann P, Ko AT, Damber JE, Logothetis C, Marberger M, Schmitz-Drager BJ, Tubaro A, Harms CJ, Roehrborn C. The VIOXX in Prostate Cancer Prevention study: cardiovascular events observed in the rofecoxib 25 mg and placebo treatment groups. Curr Med Res Opin. 2007 Sep;23(9):2063-70. doi: 10.1185/030079907X219526. PMID 17651539
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html